CLINICAL TRIAL: NCT02504606
Title: A Randomized, Open-label, Single Dose, 2-Treatment, 2-Period, 2-Way Crossover Study to Assess Safety and Pharmacokinetics of Besylsartan Tablet in Healthy Male Subject
Brief Title: Safety and Pharmacokinetics of Besylsartan Tablet in Healthy Male Subject
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Huons Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HU-009-01
Record Dates: First submitted 2015-07-17; First posted 2015-07-22 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Besylsartan (Experimental): amlodipine besylate 6.944mg+losartan K 100mg
  Interventions: Drug: Besylsartan
- Amosartan (Active Comparator): amlodipine besylate 7.841mg+losartan K 100mg
  Interventions: Drug: Amosartan

INTERVENTIONS:
Drug: Besylsartan — Amlodipin besylate 6.944mg+Losartan K 100mg
  Arms: Besylsartan
Drug: Amosartan — Amlodipin besylate 7.841mg+Losartan K 100mg
  Arms: Amosartan

SUMMARY:
This clinical trial was evaluated to compare the safety and pharmacokinetics of Besylsartan with Amosartan, which was available commercially after single oral dose in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 18 and 30
* Healthy as determined by a responsible physician

Exclusion Criteria:

* History of clinically significant disease
* Any chronic disease
* Creatine clearance less than 50ml/min
* Hypotension (100mmHg/60mmHg)
* Treatment of barbital type drug within 1 month
* Administration of herbal medicine within 7 days

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in blood concentration of Amlodipine | 144 hour
  Detect the change of blood concentration of Amlodipine by LC-MS/MS
Change from baseline in blood concentration of Losartan | 10 hour
  Detect the change of blood concentration of Losartan by LC-MS/MS